CLINICAL TRIAL: NCT05503459
Title: The Relationships Among Executive Functions, Self-regulation and Physical Exercise in Children With Autism Spectrum Disorder
Brief Title: Exercise and Cognition in Children With ASD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Education University of Hong Kong (Other)
Collaborators: San Francisco State University (Other); University of California, Riverside (Other)
Responsible Party: Principal Investigator, Andy Tse Choi-yeung, Associate Professor and Acting Head of Department, Education University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: EduUHK
Record Dates: First submitted 2022-08-11; First posted 2022-08-16 (Actual); Last update posted 2022-08-23 (Actual); Status verified 2022-08

CONDITIONS: Cognitive Impairment; Child Autism
Keywords: Cognitive function; Self-regulation; Executive Function; Physical exercise; Children; Autism
MeSH Terms: conditions — Cognitive Dysfunction; Autistic Disorder; Self-Control; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The staff responsible for the cognitive assessments and data analyses were not aware of the participants' group assignments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Bicycle learning (Experimental): The protocol for this intervention group was a 2-week bicycle training program consisting of 10 sessions (five sessions per week, 60 mins per session) in a hall/gymnasium of each participating school and the Education University of Hong Kong. Each intervention session was conducted by a professional cycling instructor assisted by student helpers. The staff-to-participant ratio was 1:1.
  Interventions: Other: Bicycle learning
- Stationary cycling group (Experimental): Participants were asked to ride on a stationary bicycle in the same format as that in the learning to bicycle group.
  Interventions: Other: Stationary cycling
- Active control group (No Intervention): Participants were asked to walk with their major caregivers for 20 minutes every day during the study period. After the study, they were taught how to ride a bicycle to recognize their contribution as controls.

INTERVENTIONS:
Other: Bicycle learning — The 10 intervention sessions were conducted in an identical format, comprising three activities: warm-up (10 min), bicycle learning (40 min), and cool-down (10 min). In the bicycle training activity, participants were asked to ride on a training bicycle with training wheels to gain better control of the bike in a gradual way. Participants then progressed from the training bicycle to a two-wheel bicycle. To keep participants on the learning curve, they were asked to ride through an obstacle course that was progressively more difficult to negotiate. The obstacles were designed by a focus group, which consisted of four physical education teachers from participating schools and one experienced cycling coach with more than five years of coaching experience.
  Arms: Bicycle learning
Other: Stationary cycling — The 10 intervention sessions were conducted in an identical format, comprising three activities: warm-up (10 min), stationary cycling (40 min), and cool-down (10 min). For stationary cycling activity, they were also asked every 10 mins during exercise to indicate their ratings of perceived exertion (target range: 3-5). Participants were positively reinforced verbally with compliments for their efforts in the training program and their daily improvements were visualized through graphs kept in the child's home.
  Arms: Stationary cycling group

SUMMARY:
Physical exercise is widely reported to be beneficial to executive functions (EFs) in children with autism spectrum disorder (ASD). However, the impact of physical exercise on self-regulation (SR) in this population remains unknown. Moreover, very few studies have been done to examine the mechanism(s) that underlie the exercise-EF and exercise-SR relationships. The purposes of the present study were to test whether two types of physical exercise (cognitively engaging vs. non-cognitively engaging) benefited SR, and if the social, emotional and physical needs of an individual mediated the exercise-EF and exercise-SR relationships. Children diagnosed with ASD were randomly assigned into one of three groups: learning to ride a bicycle (n = 23), stationary cycling (n = 19) or an active control with walking (n = 22). Two EFs (flexibility and inhibition), SR and the mediating roles of perceived social support, enjoyment, stress, physical self-efficacy and perceived physical fitness were assessed.

DETAILED DESCRIPTION:
Given the well-evidenced cognitive benefits of physical exercise for executive functions (EFs) in children with typical development (TD), there is growing research interest in whether such benefits could also be translated to children with autism spectrum disorder (ASD). Previously, the investigators examined the effectiveness of a 12-week basketball training intervention on inhibition control and working memory in children with ASD. Results showed that the training improved inhibition control. More recently, Liang and colleagues (2022) conducted a meta-analysis of seven studies examining the effect of physical exercise interventions on EFs in children and adolescents with ASD. They concluded that chronic exercise interventions were beneficial to overall EFs in the population, particularly for cognitive flexibility and inhibitory control. While physical exercise appears to be beneficial in this population, the mechanism by which physical exercise potentially impacts EFs in children with ASD remains a question. It is important to understand the mechanism in order to design an effective physical exercise intervention to promote the development of EFs among children with ASD.

Over the past few decades, most of the studies examining the exercise-cognition relation in the general population have viewed the mediating mechanism via a neurobiological framework, expressed most clearly by the neurotrophic hypothesis. The hypothesis states that physical activity increases metabolic demands and triggers a cascade of biochemical changes, such as enhancing cerebral blood blow and increasing the availability of brain-derived neurotrophic factor, which strengthens brain plasticity for higher-level cognitive activities such as those involved in executive functions. It is not until recently that scientists started questioning whether the exercise-cognition relation could also be mediated by a person's social, emotional, and physical needs. Diamond and Ling (2016) hypothesized that the most successful approaches for improving EFs would address social, emotional and physical needs, and that cognitively engaging physical activity (e.g., martial arts, dance) that enhances social interaction and joy would be more beneficial to EFs than less cognitively engaging physical activity. To the best of our knowledge, no previous studies have examined the possible mediating roles of social support, emotion and physical fitness in the exercise-EF relation.

Also of interest is the impact of physical exercise on self-regulation. Self-regulation (SR) is a psychological construct that encompasses a range of functional behaviors, such as interacting with peers, remembering rules and regulations, controlling emotions and inhibiting inappropriate and aggressive actions. Given these behaviors call upon the higher-order cognitive processes associated with EFs (e.g., shifting attention, working memory, inhibition), and the fact that SR and EFs predict many of the same positive outcomes (e.g., physical health, mental health, academic achievement), SR has long been thought of as the behavioral manifestation of EFs. However, several recent studies provided compelling evidence that SR and EFs are distinguishable and should be treated independently. Confusion may arise when measuring one without the other. Therefore, it is important to investigate whether physical exercise could yield similar benefits in SR as those in EFs, particularly in children with ASD where SR difficulties are common.

Therefore, the purposes of this study were to examine the exercise-SR relation, and to investigate the possible mediating roles of social and emotional experience and physical perception in the exercise-EF and exercise-SR relationships in children with ASD. In the present study, these needs were expressed by individuals' perceived social support, enjoyment, stress, physical self-efficacy and perceived physical fitness. Similar to our previous study, the investigators compared EFs among three groups: 1) learning to ride a bicycle, 2) stationary cycling and 3) active control (walking) before and immediately after the two-week intervention period. Following the suggestion by Diamond and Ling (2016), the active control group with walking (instead of a no-treatment control group) was used to control for potential Hawthorne effects. Walking was chosen because it was a low intensity physical activity that enabled us to assess the same potential mediators as those in the intervention groups. Unlike our previous study, only inhibition and flexibility were measured in this study because exercise interventions were shown effective to improve these two EFs in children with ASD, and to enhance the feasibility of the study (to avoid overburdening participants with the additional mediation assessments compared to our previous study). To examine the mediating effects, perceived social support, enjoyment, stress, physical self-efficacy, and perceived physical fitness were measured during the baseline period, mid-intervention and post-intervention.

ELIGIBILITY:
Inclusion Criteria:

* age 8 - 12 years
* mild to moderate ASD (i.e., level 1-2 support classification) diagnosis from physicians or psychologists based on the Diagnostic and Statistical Manual of Mental Disorders, 5th edition, (DSM-5) and Autism Diagnostic Observation Schedule, 2nd Edition (ADOS-2)
* non-verbal IQ over 50 using a brief version of the Wechsler Intelligence Scale for Children (Chinese revised) [C-WISC]
* able to follow instructions with the assistance of research staff
* able to perform the requested physical intervention, executive function measures and mediator measures with the assistance of the research staff
* no additional regular participation in physical exercise other than school physical education classes for at least one month prior to the study
* novice at riding a two-wheel bicycle (i.e., cannot ride the bicycle alone for more than 10 consecutive seconds).

Exclusion Criteria:

* other medical conditions that limited physical exercise capacities (e.g., asthma, seizure, cardiac disease)
* a complex neurologic disorder (e.g., epilepsy, phenylketonuria, fragile X syndrome, tuberous sclerosis)
* suffering from obesity (i.e., > 95 percentile of age-gender specific BMI cutoff, such that it would be difficult for research staff to catch them if they began to fall when riding
* self-reported color blindness.

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 82 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-05-28 (Actual); Study Completion 2022-06-03 (Actual)

PRIMARY OUTCOMES:
Change of cognitive flexibility | The outcome measure was conducted day 1 before intervention and within 30 minutes after intervention.
  The change of cognitive flexibility was measured by change of interference scores in the Stroop Color and Word Test between pre- and post-intervention. In the test, the participants were required to read three different tables as fast as they could. The three different tables were classified into two conditions: congruent and incongruent conditions. And the interference score was calculated based on a recognized formula ((Maximum:120; Minimum: 0). Lower interference scores indicate better cognitive flexibility.
Change of inhibition | The outcome measure was assessed day 1 before intervention and within 30 minutes after intervention.
  The change of inhibition was measured by the change of false alarm scores in the Go/No-go test between pre- and post-intervention. In this assessment, participants were asked to press a left or right key as quickly as possible when the corresponding arrow appeared on the center of a computer screen (Go response), and not to press any key whenever the up arrow appeared on the screen (No-go response). The participants completed 300 trials: 220 trials requiring a Go response (110 left and 110 right) and 80 trials (26.7%) requiring a No-go response (not pressing any key). The stimuli were randomly presented, one at a time, for 500 ms followed by 1000 ms of blank interval using E-Prime 3.0 software . After blocks of 60 trials, children were offered a break of 2 minutes. A Go response in a No-go trial was coded as a false alarm. FA errors are considered an indicator of inhibition (maximum 60; minimum: 0), and the lower the error, the better the inhibition.
Perceived social support | The outcome measure was conducted immediately after 5th intervention (day 5).
  The perceived social support of the participant was assessed with a self-reported scale referenced on the Athlete Received Support Questionnaire. Considering the comprehension difficulties of the participants, six items were chosen by the focus group (consisting of the authors, caregivers and teachers of the participants). Each participant was asked to rate their perceived social support with verbal prompting from their partnered student helpers. The total score was computed from the scale (Maximum:6; Minimum: 0). The higher the score, the better the perceived social support.
Enjoyment | The outcome measure was conducted immediately after 5th intervention (day 5).
  Participants were assisted in rating their enjoyment of the interventions and walking (active control) using the Physical Activity Enjoyment Scale. The scale was rated on 5-point Likert scale). The total score was computed from the scale (Maximum: 20; Minimum: 0). The higher the total score, the better the enjoyment.
Stress level | The outcome measure was conducted immediately after 5th intervention (day 5).
  Referenced on the Feeling Scale, a stress scale was designed by the focus group in the present study. Similar to the Feeling Scale, participants were asked to indicate their stress level from "very relaxed" (+5) to "very stressed" (-5) during the middle of the intervention. The higher the score, the lower the stress level.
Physical self-efficacy | The outcome measure was conducted immediately after 5th intervention (day 5).
  Participants were assisted in rating their self-efficacy in the interventions and walking (active control) using the Physical Self-efficacy Scale. This scale is rated on 4-point Likert scale. The total score was computed from the scale (Maximum:16; Minimum: 0). The higher the total score, the better an individual's physical self-efficacy
Perceived physical fitness | The outcome measure was conducted immediately after 5th intervention (day 5).
  Participants were asked 'How could you evaluate our own physical fitness when comparing with others?' and told to answer using a five-point scale (Maximum: 5; Minimum:0). The higher the rating, the better the perceived physical fitness.

CONTACTS AND LOCATIONS:
Locations (1):
- EdUHK, Hong Kong, China, Hong Kong

IPD SHARING:
Plan to Share IPD: No